CLINICAL TRIAL: NCT02530268
Title: Corrona Psoriatic Arthritis and Spondyloarthritis (PsA-SpA) Registry
Brief Title: The Corrona Psoriatic Arthritis and Spondyloarthritis (PsA-SpA) Registry
Status: Enrolling by invitation | Type: Observational
Sponsor: CorEvitas (Network)
Responsible Party: Sponsor
Other Study IDs: Corrona-PSA-400
Record Dates: First submitted 2015-05-01; First posted 2015-08-21 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Psoriatic Arthritis; Spondyloarthritis
Keywords: psoriatic arthritis; spondyloarthritis; disease registry
MeSH Terms: conditions — Arthritis, Psoriatic; Spondylarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ankylosing Spondylitis: Pts presenting to enrolling sites across the US are invited to enroll if eligible
- Psoriatic Arthritis: Pts presenting to enrolling sites across the US are invited to enroll if eligible

SUMMARY:
This prospective, non-interventional, research registry is designed to study the comparative effectiveness and comparative safety of approved treatments for PsA-SpA in a cohort of patients cared for by rheumatologists across North America. Secondary objectives include analyzing the epidemiology and natural history of the disease, its comorbidities, and current treatment practices.

DETAILED DESCRIPTION:
There is a significant unmet need to develop clinical registry data on the presentation, natural history, management, and outcomes of PsA-SpA. There is no large clinical registry of PsA-SpA patients seen in general rheumatology practices. It is anticipated that Corrona's registry will supplement information gathered in other programs and potentially represent a more general rheumatology spectrum of PsA-SpA patients representative of the general population.

The primary objective of the registry is to prospectively study the comparative effectiveness and comparative safety of therapies in a national cohort of PsA-SpA patients being cared for by rheumatologists. Secondary objectives include analyzing the epidemiology and natural history of the disease group, comorbidities, and current treatment practices.

The design is a prospective, non-interventional, observational registry for patients with PsA or SpA under the care of a licensed rheumatologist. Longitudinal follow-up data is collected from both patients and their treating rheumatologists during routine clinical encounters using Corrona registry questionnaires. These questionnaires collect data on patient demographics, disease duration, medical history (including all prior and current treatments for PsA-SpA), smoking status, alcohol use, disease severity, pain, activity, and other clinical effectiveness measures, patient reported outcomes, comorbidities, hospitalizations, and other targeted safety outcomes, including pregnancy.

After the enrollment visit, SpA patients and physicians will complete follow-up questionnaires during regularly scheduled clinical encounters. The goal is to collect data from patients and providers at six month intervals, not to exceed 2 visits in any 12 month period.

Adverse events may be volunteered spontaneously by the subject, or be discovered as a result of general questioning by the Principal Investigator. During all Corrona related visits with the Principal Investigator, subjects will be questioned regarding the occurrence of adverse events.

ELIGIBILITY:
To be eligible for enrollment into the Corrona PsA-SpA Registry, a patient must satisfy all of the inclusion criteria and none of the exclusion criteria listed below.

Inclusion Criteria

The patient must be:

1. One of the following:

   1. Diagnosed with psoriatic arthritis (PsA) and initiating (prescribed or starting) an eligible medication† for the treatment of PsA at the enrollment visit.
   2. Meet the ASAS criteria for axial spondyloarthritis (AxSpA), including radiographic or non-radiographic, and initiating (prescribed or starting) an eligible biologic for the treatment of AxSpA at the enrollment visit.
   3. Meet the modified New York classification criteria for ankylosing spondylitis (AS) and initiating (prescribed or starting) an eligible biologic for the treatment of AS at the enrollment visit
2. At least 18 years of age or older
3. Able and willing to provide written consent

Exclusion Criteria

The patient must not be:

1. Diagnosed with rheumatoid arthritis, systemic lupus erythematosus, or any other form of autoimmune inflammatory arthritis.
2. Participating in or planning to participate in a clinical trial with an interventional research study of a non-marketed or marketed investigational drug (e.g. phase I-IV clinical drug trial, post marketing study or registry study where drug is being provided). Of note, concurrent participation in another observational registry study is not excluded. ∆

   * Once clinical trial participation has ended, a patient is permitted to enroll in the registry if they satisfy the eligibility requirements at the time of enrollment. If the patient participated in the PsA-SpA registry and was exited to join a clinical trial, the patient cannot be re-enrolled in the PsA-SpA registry after clinical trial participation has ended.

Patients switching from an originator biologic to a biosimilar satisfy the enrollment eligibility requirement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are enrolled in the Psoriatic Arthritis and Spondyloarthritis Registry during regularly scheduled office visits. Selected rheumatologists are invited to participate as investigators in the Registry.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2013-03; Primary Completion 2100-12 (Estimated); Study Completion 2100-12 (Estimated)

PRIMARY OUTCOMES:
The major clinical outcomes include an assessment of the epidemiology of Spondyloarthritis; to better understand the presentation, natural history, management and outcomes. | A minimum of 10 years from last patient enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Greenberg, MD, MPH, Study Director — CorEvitas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mease PJ, Blachley T, Malatestinic WN, Harrold LR, Dube B, Lisse JR, Bolce RJ, Hunter TM. Effectiveness of bDMARDs in ankylosing spondylitis patients by biologic use: experience from the CorEvitas PsA/SpA Registry. Curr Med Res Opin. 2024 Feb;40(2):315-323. doi: 10.1080/03007995.2023.2291160. Epub 2024 Jan 24. PMID 38050693
- [Derived] Mease PJ, Ogdie A, Tesser J, Shiff NJ, Lin I, Chakravarty SD, Kelleman M, Dodge R, McLean RR, Broadwell A, Kavanaugh A, Merola JF. Six-Month Persistence and Multi-domain Effectiveness of Guselkumab in Adults with Psoriatic Arthritis: Real-World Data from the CorEvitas Psoriatic Arthritis/Spondyloarthritis Registry. Rheumatol Ther. 2023 Dec;10(6):1479-1501. doi: 10.1007/s40744-023-00582-w. Epub 2023 Aug 19. PMID 37597159
- [Derived] Mease PJ, Accortt NA, Rebello S, Etzel CJ, Harrison RW, Aras GA, Gharaibeh MMF, Greenberg JD, Collier DH. Persistence of tumor necrosis factor inhibitor or conventional synthetic disease-modifying antirheumatic drug monotherapy or combination therapy in psoriatic arthritis in a real-world setting. Rheumatol Int. 2019 Sep;39(9):1547-1558. doi: 10.1007/s00296-019-04345-1. Epub 2019 Jul 18. PMID 31321485
- See also: CorEvitas home page — https://www.corevitas.com/